CLINICAL TRIAL: NCT00807222
Title: Study of the Effect of Vyvanse (Lisdexamfetamine Dimesylate) on Sleep in Children Aged 6-12 Years With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Effect of Vyvanse on Sleep in Children Aged 6-12 Years With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Study Centers, LLC (Other)
Collaborators: Shire (Industry)
Responsible Party: John Martin Giblin, MD / President/CEO, Medical Director, Clinical Study Centers, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IST-NRP104
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Sleep
Keywords: ADHD; Vyvanse; lisdexamfetamine dimesylate; LDX; sleep
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lisdexamfetamine dimesylate (Active Comparator): 30, 50, or 70 mg
  Interventions: Drug: lisdexamfetamine dimesylate
- placebo (Placebo Comparator)
  Interventions: Drug: lisdexamfetamine dimesylate

INTERVENTIONS:
Drug: lisdexamfetamine dimesylate — Subjects will receive Vyvanse 30, 50, or 70 mg per day or placebo capsules orally for up to (a maximum of) seven (7) weeks.
  Other Names: Vyvanse

SUMMARY:
This study involves research to test how Vyvanse (study drug) affects sleep in 24 children aged 6 to 12 years who have ADHD. Vyvanse is approved by the FDA for the treatment ADHD of in children aged 6 to 12 years. The experimental part of this study is to determine how Vyvanse affects sleep.

DETAILED DESCRIPTION:
Treatment with psychostimulants has been associated with sleep disturbances, including both sleep onset and maintenance problems, in children with ADHD. This analysis evaluated the effect of lisdexamfetamine dimesylate (LDX) on sleep in children with ADHD.

This single center, double-blind, placebo-controlled, parallel-group trial enrolled children aged 6-12 years with a DSM-IV-TR diagnosis of ADHD. The study included a screening period, 1-week washout, 3-week open-label LDX dose optimization phase, and a 4-week double-blind treatment phase in which subjects were randomized to placebo or active LDX treatment at 30, 50, or 70 mg/d. Polysomnograph and actigraph measures as well as assessments of subjective sleep parameters were performed in all subjects prior to treatment and reassessed after treatment with either LDX or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject 6 to 12 years of age, inclusive
2. Subject meets DSM-IV-TR criteria for a primary diagnosis of ADHD
3. Female subjects of childbearing potential (FOCP) must have a negative urine pregnancy test
4. Subject must be in general good health
5. Subject's parent or legally authorized guardian provides signature of informed consent, and there is documentation of assent by the subject.
6. Subject and parent/caregiver are willing and able to comply with all the testing and requirements defined in the protocol.
7. Subject is generally functioning academically at age-appropriate levels
8. Subject is able to swallow a capsule.
9. Subject and parent/guardian are willing to comply with entire visit schedule for the study and Sleep Hygiene Instructions

Exclusion Criteria:

1. Subject has a comorbid psychiatric diagnosis that contraindicates VyvanseTM treatment or would confound efficacy or safety assessments.
2. Subject has any comorbid illness that could interfere with participation in the study.
3. Subject is a known non-responder to an adequate trial of stimulant medication for ADHD.
4. Subject has history of symptoms or has an identified sleep disorder
5. Subject has a history of seizure during the last 2 years
6. Subject is significantly overweight or obese
7. Subject has any clinically significant ECG or laboratory abnormalities at screening or baseline.
8. Subject has any specific cardiac condition or family history of cardiac disease
9. Subject is taking medications that affect blood pressure or heart rate (except current ADHD therapy, if any).
10. Subject has a positive urine drug result at screening (except current ADHD therapy, if any).
11. Subject is hypertensive.
12. Subject has any documented adverse reactions, allergy, or intolerance to amphetamines or dextroamphetamines.
13. Subject is taking exclusionary medications
14. Subject currently has (or had a history in the previous 12 months) a drug dependence or substance abuse disorder
15. Subject has taken another investigational product or taken part in a clinical trial within the 30 days prior to Screening (Visit 1).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Latency to Persistent Sleep (LPS) as measured by polysomnography (PSG) | performed at Baseline (Visit 2), after the subject has met all other inclusion/exclusion criteria, and at Week 7 or Early Termination

SECONDARY OUTCOMES:
PSG sleep parameters: Wake time After Sleep Onset (WASO), Number of Awakenings After Sleep Onset (NAASO), and Total Sleep Time (TST) | within four days prior to Baseline (Visit 2), after the subject has met all other inclusion/exclusion criteria and Week 7 or Early Termination (Visit 9)
Actigraphic measures of sleep characteristics (LPS, TST) | during the week immediately preceding the following study visits: Visit 2 (Baseline), Visit 5 (Week 3), and Visit 9 (Week 7)
Pittsburgh Sleep Quality Index and Child Sleep Habits Questionnaire item scores | performed at Visits 2 through 9
Clinical Global Impression (CGI) Severity and Global Improvement item scores | each weekly visit
Conner's Parent Rating Scale - Revised (S) completed by parent/caregiver and Investigator-rated ADHD-RS-IV item scores | Visits 2 through 9

CONTACTS AND LOCATIONS:
Overall Officials: John M Giblin, MD, Principal Investigator — Clinical Study Centers, LLC
Locations (1):
- Clinical Study Centers, LLC, Little Rock, Arkansas, United States